CLINICAL TRIAL: NCT06835686
Title: LA-CEAL CONNECT: Louisiana Community Engagement Alliance (LA-CEAL) Collaborative Multi-level Obesity Intervention Engaging Underserved Communities Trial (CONNECT)
Brief Title: Collaborative Multi-level Obesity Intervention Engaging Underserved Communities Trial
Acronym: CONNECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-822; OT2HL158287 (NIH)
Record Dates: First submitted 2025-01-12; First posted 2025-02-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Health Literacy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LA-CEAL CONNECT Intervention (Experimental): Participants will receive: 1) culturally tailored and health literacy-appropriate educational materials about weight loss and obesity, 2) health coaching from community health workers over 6 months, and 3) digital weight scale and fitness tracker (e.g., Fitbit).
  Communities will receive support to conduct Community Asset Mapping and design and implement Community Action Projects to promote health resources in their community.
  FQHC clinic providers will receive: 1) education on guideline-based obesity management, 2) toolkit with resources for obesity management.
  Interventions: Behavioral: Health Literacy and Culturally Tailored Materials; Behavioral: Community-Engaged Health Coaching and Navigation; Behavioral: Self-Monitoring and Remote Patient Monitoring of weight and physical activity; Other: Community Asset Mapping (CAM); Other: Primary Care Provider Training; Other: Obesity Toolkit for Primary Care Providers
- Enhanced Usual Care (Active Comparator): Participants will receive culturally tailored and health literacy-appropriate educational materials about weight loss and obesity. FQHC clinic providers will receive education on obesity management.
  Interventions: Behavioral: Health Literacy and Culturally Tailored Materials; Other: Primary Care Provider Training

INTERVENTIONS:
Behavioral: Health Literacy and Culturally Tailored Materials — Participants will receive health literacy-appropriate written information on community resources and weight management
Behavioral: Community-Engaged Health Coaching and Navigation — Participants will receive virtual coaching sessions over a 6-month period from trained Community Health Workers (CHWs). Coaching will include culturally competent information and strategies for weight management, and linking participants to community wellness resources identified in Community Asset Mapping (see below). Coaches will also remotely monitor patients' weight loss and physical activity via online portals to provide patients with tailored support during coaching sessions.
  Arms: LA-CEAL CONNECT Intervention
Behavioral: Self-Monitoring and Remote Patient Monitoring of weight and physical activity — Participants will self-monitor weight and physical activity during the 6-month health coaching protocol using a cellular-connected digital weight scale and a Bluetooth-connected wrist-worn fitness tracking device (e.g., Fitbit). Participants will be instructed to weigh themselves and wear a fitness tracker (e.g., Fitbit) daily. Health coaches will remotely monitor weight and physical activity data logged by these devices to incorporate into health coaching sessions.
  Arms: LA-CEAL CONNECT Intervention
Other: Community Asset Mapping (CAM) — The CHW from each intervention community clinic will convene a team of community members, including but not limited to CONNECT participants, that will meet regularly to identify and describe community assets that enable, support, and promote healthy lifestyles related to weight loss and management (e.g., healthy eating and physical activity resources). Community teams will be supported to design and implement Community Action Projects to promote the utilization of community resources identified in the map.
  Arms: LA-CEAL CONNECT Intervention
Other: Primary Care Provider Training — Education sessions will be provided to FQHC providers. The training curriculum is designed to increase healthcare providers' knowledge of evidence-based and guideline-concordant obesity management strategies in primary care settings.
Other: Obesity Toolkit for Primary Care Providers — We will provide FQHC providers with a toolkit containing additional obesity management resources and information and the community resource guides given to participants to support obesity management.
  Arms: LA-CEAL CONNECT Intervention

SUMMARY:
The goal of this clinical trial is to test the effectiveness of an evidence-based multi-level intervention for weight loss and the feasibility, fidelity, and sustainability of implementing the intervention in low-income and underserved people living with obesity in Louisiana. The main questions it aims to answer are:

* Will an evidence-based multi-level obesity intervention (called LA-CEAL CONNECT) in adults living with obesity in low-income and underserved communities achieve weight loss at 6 months compared to enhanced usual care?
* Will LA-CEAL CONNECT sustain weight loss at 12 months?
* Will LA-CEAL CONNECT improve waist circumference, diet quality, physical activity, quality of life, and blood pressure at 6 and 12 months?
* Will LA-CEAL CONNECT be feasible to implement in adults living with obesity in low-income and underserved communities?

Researchers will compare the LA-CEAL CONNECT multilevel weight loss intervention to enhanced usual care to evaluate if LA-CEAL CONNECT leads to greater weight loss and greater changes in waist circumference, diet, physical activity, quality of life, and blood pressure than enhanced usual care.

Participants in both arms will:

* Receive health literacy-tailored educational materials and resources for weight loss
* Visit the clinic site for baseline, 6-month and 12-month study visits to collect clinical and survey measurements

Participants in the CONNECT intervention arm will also:

* receive health coaching
* self-monitor weight and physical activity using digital technologies
* attend group meetings to identify and increase utilization of community health and wellness resources

ELIGIBILITY:
Inclusion Criteria:

* being 18 to 75 years of age
* living with obesity, defined as a BMI between 30 and 50 kg/m2 for non-Asian identifying participants and BMI between 27.5 and 50 kg/m2 for Asian-identifying participants
* weighing less than 400 pounds
* receiving care from or willing to register at a participating FQHC clinic
* able to understand and speak English
* able to complete the study within the next year (e.g., not planning to move from the area within study period)

Exclusion Criteria:

* having given birth within the past year, pregnant or planning to become pregnant during study period (within 1 year)
* currently participating in a weight-loss program
* having lost more than 10 pounds in the last 6 months
* being an employee or a family member of an employee of any participating FQHC
* having a disease that can interfere with or be aggravated by exercise or weight loss

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in % weight change | 6 months
  Trained personnel will measure weight at all visits using a digital weight scale. For weight, measurement will be performed twice, with a third measurement if the first 2 measurements deviate more than 0.1 kg. An average of the two closest measurements will be used for analyses.

SECONDARY OUTCOMES:
Between-group difference in change in waist circumference | 6 months
  Trained personnel will measure waist circumference at all study visits using a non-elastic tape measure placed on the skin in a horizontal plane around the abdomen at the level of the iliac crest. The measurement will be performed twice, with a third measurement if the first 2 measurements deviate more than 0.5 cm; average of the two closest measurements will be used for analyses.
Between-group difference in change in blood pressure | 6 months
  Systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be measured at every study visit using an oscillometric Omron Professional Intellisense Blood Pressure Monitor HEM-907XL and following the American Heart Association (AHA) protocol.
Between-group difference in change in dietary intake | 6 months
  Diet will be self-reported at every study visit using a diet screener that has been developed by the study investigators and used in past studies. The screener will assess frequency of consumption of selected food and drinks over the past month - including fruits and vegetables, high-fat foods, and alcoholic beverages.
Between-group difference in change in physical activity | 6 months
  Physical activity will be self-reported at every study visit using the 7-item international physical activity questionnaire - short form (IPAQ-SF). This tool records the time spent at 4 different activity levels (vigorous, moderate, walking, sitting) according to 7-day recall. Scores are computed by calculating total minutes/week or total MET-minutes/week spent in the following activity levels: vigorous, moderate, walking, sitting. A total physical activity score is computed by summing the values for vigorous, moderate, and walking domains. The minimum score is 0 (no activity), with higher scores indicating more physical activity. The categorical physical activity level (low, moderate, and high) will be calculated using cut points recommended by the authors. Continuous activity score may be used as a more sensitive measure of participant physical activity change.
Between-group difference in change in quality of life | 6 months
  Quality of life will be self-reported at every study visit using the 10-item Patient Reported Outcomes Measurement Information System (PROMIS) Global Health measure. Raw scores for Global Physical Health and Global Mental health will be computed, ranging from 4 to 20. Per PROMIS scoring guidelines, raw scores will be transformed to a T-score metric, with higher scores representing better health on each domain.

OTHER OUTCOMES:
Between-group difference in % weight change | 12 months
  Change in weight from the baseline visit to the 12 month visit using a standard protocol (see above).
Between-group difference in change in waist circumference | 12 months
  Change in waist circumference from the baseline visit to the 12 month visit using a standard protocol (see above).
Between-group difference in change in blood pressure | 12 months
  Change in SBP and DBP from baseline visit to 12 month visit using a standard protocol (see above).
Between-group difference in change in dietary intake | 12 months
  Diet will be self-reported at every study visit using a diet screener that has been developed by the study investigators and used in past studies. The screener will assess frequency of consumption of selected food and drinks over the past month - including fruits and vegetables, high-fat foods, and alcoholic beverages.
Between-group difference in change in physical activity | 12 months
  Physical activity will be self-reported at every study visit using the 7-item international physical activity questionnaire - short form (IPAQ-SF). This tool records the time spent at 4 different activity levels (vigorous, moderate, walking, sitting) according to 7-day recall. Scores are computed by calculating total minutes/week or total MET-minutes/week spent in the following activity levels: vigorous, moderate, walking, sitting. A total physical activity score is computed by summing the values for vigorous, moderate, and walking domains. The minimum score is 0 (no activity), with higher scores indicating more physical activity. The categorical physical activity level (low, moderate, and high) will be calculated using cut points recommended by the authors. Continuous activity score may be used as a more sensitive measure of participant physical activity change.
Between-group difference in change in quality of life | 12 months
  Quality of life will be self-reported at every study visit using the 10-item Patient Reported Outcomes Measurement Information System (PROMIS) Global Health measure. Raw scores for Global Physical Health and Global Mental health will be computed, ranging from 4 to 20. Per PROMIS scoring guidelines, raw scores will be transformed to a T-score metric, with higher scores representing better health on each domain.
Between-group difference in fidelity | 6 months
  Composite measure of fidelity comprised of self-reported frequency of weight measurement, receipt of health coaching, and use of community resources that support healthy lifestyles.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Krousel-Wood, MD, MSPH, Principal Investigator — Tulane University
Locations (18):
- United States (18):
  - InclusivCare - Avondale Clinic, Avondale, Louisiana
  - CommuniHealth Services - Bastrop Clinic, Bastrop, Louisiana
  - CareSouth Medical and Dental - Baton Rouge Clinic, Baton Rouge, Louisiana
  - Teche Action Clinic - Franklin, Franklin, Louisiana
  - Southeast Community Health Systems - Greensburg Clinic, Greensburg, Louisiana
  - Teche Action Clinic - Houma, Houma, Louisiana
  - Southeast Community Health Systems - Independence Clinic, Independence, Louisiana
  - InclusivCare - Kenner Clinic, Kenner, Louisiana
  - RKM Primary Care - Loranger Clinic, Loranger, Louisiana
  - InclusivCare - Marrero, Marrero, Louisiana
  - David Raines Community Health Center - Minden Clinic, Minden, Louisiana
  - Teche Action Clinic - Morgan City, Morgan City, Louisiana
  - NOELA Community Health Center, New Orleans, Louisiana
  - Teche Action Clinic - South Pierre Part, Pierre Part, Louisiana
  - CareSouth Medical and Dental - Plaquemine Clinic, Plaquemine, Louisiana
  - David Raines Community Health Center - Shreveport Clinic, Shreveport, Louisiana
  - RKM Primary Care - Springfield Clinic, Springfield, Louisiana
  - CommuniHealth Services - West Monroe Clinic, West Monroe, Louisiana